CLINICAL TRIAL: NCT07374055
Title: Effects of the Geriatric Nutritional Risk Index (GNRI), Mini Nutritional Assessment-Short Form (mNA-SF), and Systemic Immune-Inflammation Index (SII) on Postoperative Morbidity and Mortality in Geriatric Patients Undergoing Gastrointestinal Surgery
Brief Title: The Effect of Nutritional Status on Postoperative Mortality and Morbidity in the Geriatric Population Undergoing Gastrointestinal Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Minel Neslihan, Assistant Doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: KARTALANESTEZİ088
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Nutrition Assessment; Geriatric Anesthesia
Keywords: Geriatric; Nutritional; Mortality; Gastrointestinal surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Gastrointestinal Surgery Patients.: This group consists of 200 geriatric patients aged 65 and older who are scheduled to undergo gastrointestinal surgery. Participants are within the ASA 3-4 risk groups and must have a Mini-Mental State Examination (MMSE) score of 21 or higher to be included.
  Interventions: Other: Preoperative Risk Scoring; Other: Postoperative Morbidite and Mortality Monitoring; Other: Delirium Assessment Protocol

INTERVENTIONS:
Other: Preoperative Risk Scoring — Patients will be evaluated preoperatively using three distinct scoring systems: the Geriatric Nutritional Risk Index (GNRI), the Mini Nutritional Assessment-Short Form (mNA-SF), and the Systemic Immune-Inflammation Index (SII). These scores are calculated based on serum albumin levels, body weight, a 6-question survey, and laboratory values (platelets, neutrophils, and lymphocytes).
Other: Postoperative Morbidite and Mortality Monitoring — Systematic tracking of postoperative outcomes including hospital and ICU stay duration, pulmonary complications (e.g., pneumonia, embolism), extrapulmonary complications (e.g., surgical site infection, organ failure, delirium), and mortality rates at 30, 60, and 90 days.
Other: Delirium Assessment Protocol — Patients will be monitored for delirium preoperatively, on the first postoperative day, and before discharge using the Confusion Assessment Method (CAM/CAM-ICU) and the Richmond Agitation-Sedation Scale (RASS).

SUMMARY:
The purpose of this study was to compare the sensitivity and specificity of the Geriatric Nutritional Risk Index (GNRI), Mini Nutritional Assessment Scale-Short Form (mNA-SF) and Systemic Immune-Inflammatory Index (SII) values calculated in the preoperative evaluation in patients over 65 years of age who underwent gastrointestinal surgery, in predicting morbidity and mortality in the postoperative period.

DETAILED DESCRIPTION:
It is crucial to evaluate the impact of nutritional status and systemic inflammation markers on postoperative outcomes in geriatric patients undergoing gastrointestinal surgery.

Nutritional status has a decisive impact on the development of morbidity and mortality in geriatric patients. The risk of malnutrition is particularly high in the geriatric patient population undergoing gastrointestinal surgery. Predicting postoperative outcomes in these patient groups is becoming increasingly important. To this end, many different risk scoring systems have been developed.

Low nutritional scores and increased inflammatory responses are associated with high mortality, prolonged hospitalization and intensive care unit stays, and complications. The primary goal of preoperative risk scoring is to predict potential complications before, during, and after surgery, and to minimize risks and mortality by attempting to prevent them.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo gastrointestinal surgery.

Age 65 years and older.

ASA (American Society of Anesthesiologists) physical status class 3 or 4.

Mini-Mental State Examination (MMSE) score of 21 or higher

Exclusion Criteria:

* Patients who do not consent to participate in the study.

Patients with acute infection during the preoperative period.

Patients who received albumin replacement in the preoperative period.

Patients with a Mini-Mental State Examination (MMSE) score below 21.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric patients scheduled for gastrointestinal surgery at a single-center tertiary care urban hospital (SBÜ Kartal Dr. Lütfi Kırdar City Hospital).".
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Systemic Immune-Inflammation Index (SII) | Preoperative (Baseline)
  Calculated as (Platelets x Neutrophils) / Lymphocytes from preoperative blood samples.The unit of measure is cells per microliter.
Geriatric Nutritional Risk Index (GNRI) as a predictor of postoperative complications | Preoperative (Baseline)
  GNRI will be calculated using serum albumin and body weight. Scores will be used to categorize patients' nutritional risk.Units on a scale of 0 to 120, where lower scores indicate higher nutritional risk.
Mini Nutritional Assessment-Short Form (mNA-SF) score | Preoperative (Baseline)
  A 6-question survey to screen for malnutrition.Measured on a scale of 0 to 14 points, where 0-7 indicates malnourishment.

SECONDARY OUTCOMES:
Postoperative Morbidity | Up to 30 days post-surgery
  Monitoring of pulmonary (e.g., pneumonia, embolism) and extrapulmonary (e.g., surgical site infection, organ failure, anastomosis leak) complications
Incidence of Delirium | Preoperative to discharge
  Assessment of delirium using the Confusion Assessment Method (CAM/CAM-ICU) and Richmond Agitation-Sedation Scale (RASS).
Length of Hospital and ICU Stay | Total duration of hospitalization
  Recording the number of days spent in the hospital and intensive care unit.
Postoperative Mortality Rate | 30, 60, and 90 days post-surgery
  Tracking patient survival rates at specified intervals after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Minel N KUTUPOGLU SEZER, MD, Principal Investigator — University of Health Sciences, Kartal Dr. Lutfi Kirdar City Hospital
Locations (1):
- Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.